CLINICAL TRIAL: NCT00781157
Title: Up-down Determination of the ED90 of Phenylephrine for Spinal Induced Hypotension in Parturients Undergoing Cesarean Delivery
Brief Title: Phenylephrine for Spinal Induced Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWK-4061-2007; IWK REB 4061
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Hypotension
Keywords: Spinal induced hypotension in cesarean delivery
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Phenylephrine bolus

INTERVENTIONS:
Drug: Phenylephrine bolus — The initial dose of phenylephrine will be 100 mcg, a dose within the clinical range currently in use at our center. The subsequent dose is based upon the response of the preceding subject in the usual up-and-down method (UDM), which is outlined in the "data analysis" section of the protocol. The dosing changes will be in increments of 20 micrograms. A successful response to this dose will be entered into a spreadsheet, designed by our statistician, which will determine the subsequent dose based upon the UDM. If a failure is observed in the previous subject, the dose is stepped up in the next subject. If a success is observed the next subject is randomized with probability of 0.10 to the next lower dose and with probability 0.90 to the same dose.

SUMMARY:
This study is designed to determine the ED90 for a single dose of phenylephrine for the treatment of spinal induced hypotension in parturients presenting for an elective CD. The ED90 is the effective dose at which 90% of subjects will have a "positive" response to phenylephrine. The primary outcome measure is the ED90 for bolus phenylephrine. Secondary outcomes include the need for additional vasopressors, glycopyrolate to treat bradycardia, and the presence of hypertension following administration of phenylephrine.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent cesarean delivery with planned regional anesthesia (i.e. elective planned cesarean delivery for malposition, patient choice, cervical pelvic disproportion, previous cesarean delivery and other diagnosis that require a predetermined cesarean delivery)
2. American Society of Anesthesia physical status class I & II (ASA I - Healthy, ASA II - mild and controlled systemic disease, eg. controlled essential hypertension)
3. Age ≥ 18 years (Standard within the obstetrical literature)
4. Term gestational age
5. English-speaking

Exclusion Criteria:

1. Morbid Obesity (Body Mass Index ≥ 45 kg/m2) (Morbidly obese parturients require a dose of local anesthetic less than the standardized dose in this study, typically have an exaggerated response to vasopressors, and the blood pressure cuff occasionally needs to be replaced by an intraarterial catheter due to limitations in size)
2. Height < 5'0" (Women < 5'0" are likely to require a dose of local anesthetic less than the standardized dose in this study)
3. Laboring women
4. Urgent or emergency cesarean delivery
5. Severe hypertensive disease of pregnancy defined as systolic blood pressure (SBP) > 160mmHg, diastolic blood pressure (DBP) > 110mmHg and/or requiring antihypertensive treatment or associated with significant proteinuria
6. Severe maternal cardiac disease
7. Diabetes type I
8. Subjects on monoamine oxidase inhibitors (MAOI's) or tricyclic antidepressants
9. Fetal anomalies
10. Failed spinal anesthesia
11. Subject enrollment in another study involving a study medication within 30 days of CD
12. Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the ED90 for bolus phenylephrine. | Intraoperative

SECONDARY OUTCOMES:
Secondary outcomes include the need for additional vasopressors, glycopyrolate to treat bradycardia, and the presence of hypertension following administration of phenylephrine. | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada